CLINICAL TRIAL: NCT00159068
Title: Genetic Influences on the Course and Response to Treatment of HIV: Contribution of Polymorphisms in Drug Metabolism and Disposition Genes and Haptoglobin Polymorphisms
Brief Title: Analysis of Genetic Factors Which May Influence the Course of HIV Infection
Status: Completed | Type: Observational
Sponsor: Deborah Rund (Other)
Responsible Party: Sponsor-Investigator, Deborah Rund, Senior Hematologist, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Other Study IDs: 391200-HMO-CTIL
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA isolated from peripheral blood.
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with HIV an have a variable course of their infection. We are trying to identify factors which worsen or ameliorate the course of the disease. Such factors may be related to metabolism (breakdown) of drugs or to iron handling by the body.

DETAILED DESCRIPTION:
Patients with HIV can have a variable course and the disease may be influenced by polymorphisms in drug metabolism and disposition genes such as MDR1 and CYP3A4. In addition, reports have linked changes in the course of the disease with iron status, with high iron being detrimental. We will study polymorphisms in these genes and correlate with clinical course in HIV patients and also with phenotype of drug resistance and disease parameters (such as CD4 counts and opportunistic infections).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HIV

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HIV attending the HIV clinic at Hadassah colden globes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Rund, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Tang J, Kaslow RA. The impact of host genetics on HIV infection and disease progression in the era of highly active antiretroviral therapy. AIDS. 2003;17 Suppl 4:S51-60. doi: 10.1097/00002030-200317004-00006. No abstract available. PMID 15080180